CLINICAL TRIAL: NCT04631627
Title: A Prospective Muti-center Study of Early Prediction and Randomised Prevention of Preeclampsia With Low Dose Aspirin in Chinese Cohort
Brief Title: Early Prediction and Randomised Prevention of Preeclampsia With Low Dose Aspirin in Chinese Cohort
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EPRPLACC
Record Dates: First submitted 2020-11-07; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Preeclampsia
Keywords: preeclampsia; aspirin; prediction; intervention; PAPP-A; PIGF; sFlt
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspirin group (Active Comparator): aspirin,tablet,100/150mg per day,(BMI<30 100mg/d，BMI≥30 150mg/d)，from pregnancy weeks<16 to 35 weeks or the day of delivery.
  Interventions: Drug: Aspirin
- control group (Sham Comparator): with no intervention
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — With the result of risk assessment for high risk and the risk of pregnant women, with each research center stratified random aspirin drug intervention, for each center screening high-risk and accord with the standard drug intervention study phase into eliminate pregnant women by using stochastic indicator 1:1 randomly into low-dose aspirin to prevent group and observation group, for each center in screening for risk and comply with the drug intervention study phase into the exclusion standard 1:1 by random indicator method pregnant women randomly into low-dose aspirin to prevent group and observation group.

SUMMARY:
This study intends to adopt the method of multi-center prospective randomized controlled study. The aim of this study is to obtain localized excision values through a preeclampsia screening model established in early pregnancy, and to evaluate the efficacy of low-dose aspirin intervention for preeclampsia prevention in pregnant women at high risk of screening.

ELIGIBILITY:
Inclusion Criteria:

* 1)Pregnant women assessed as at high risk of preeclampsia 2) live pregnancy 3) gestational weeks < 16 weeks 4) agree to randomized drug intervention studies 5) follow up regularly and obtain reliable pregnancy outcomes

Exclusion Criteria:

* 1)with severe fetal or chromosomal abnormalities 2) induced labor or spontaneous abortion due to social factors 3) absolute or relative contraindications to aspirin use (allergy to aspirin or other salicylate, or other ingredients of the drug;Acute gastrointestinal ulcer;Active bleeding;In patients with severe G6PD deficiency, acetylsalicylic acid may induce hemolysis or hemolytic anemia.Aspirin asthma)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — gestational women
Enrollment: 1500 (Estimated)
Dates: Start 2020-11-16 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
the rate of preeclampsia | through study completion, an average of 1 year
  Hypertensive onset after 20 weeks of gestation is accompanied by proteinuria,or with thrombocytopenia, impaired liver function, renal insufficiency,pulmonary edema,headache without other explanation and so on.
the rate of hypertensive disorder during pregnancy | through study completion, an average of 1 year
  gestational hypertension, preeclampsia, chronic hypertension with preeclampsia, eclampsia, HELLP syndrome
the rate of placenta abruption | through study completion, an average of 1 year
  After 20 weeks of pregnancy, the placenta in its normal position is completely or partially removed from the uterine wall before delivery of the fetus
the rate of fetal growth restriction | through study completion, an average of 1 year
  The birth weight of the fetus is below two standard deviations of the average weight for the same gestational age or below the 10th percentile of normal weight for the same age
the rate of postpartum hemorrhage | within 24 hours after the delivery
  Within 24 hours after the delivery of the fetus, the bleeding volume of vaginal delivery ≥500ml, cesarean delivery ≥1000ml
the time and type of delivery | within 24 hours after the delivery
  gestational week, vaginal delivery and cesarean section

SECONDARY OUTCOMES:
birth weight of newborn | delivery time
  macrosomia, normal weight, low birth weight
Apgar score for newborns | delivery time
  ≥8；4-7,；≤3
the rate of Neonatal NICU occupancy rate | through study completion, an average of 1 year
  the day of NICU occupancy

IPD SHARING:
Plan to Share IPD: Yes
The aim of this study was to obtain localized excision values through a preeclampsia screening model established in early pregnancy, and to evaluate the efficacy of low-dose aspirin intervention for preeclampsia prevention in pregnant women at high risk of screening.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 31 June, 2022

REFERENCES:
- [Background] Duley L. The global impact of pre-eclampsia and eclampsia. Semin Perinatol. 2009 Jun;33(3):130-7. doi: 10.1053/j.semperi.2009.02.010. PMID 19464502
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Akolekar R, Syngelaki A, Poon L, Wright D, Nicolaides KH. Competing risks model in early screening for preeclampsia by biophysical and biochemical markers. Fetal Diagn Ther. 2013;33(1):8-15. doi: 10.1159/000341264. Epub 2012 Aug 16. PMID 22906914
- [Background] Park F, Russo K, Williams P, Pelosi M, Puddephatt R, Walter M, Leung C, Saaid R, Rawashdeh H, Ogle R, Hyett J. Prediction and prevention of early-onset pre-eclampsia: impact of aspirin after first-trimester screening. Ultrasound Obstet Gynecol. 2015 Oct;46(4):419-23. doi: 10.1002/uog.14819. Epub 2015 Aug 31. PMID 25678383
- [Background] Sentilhes L, Azria E, Schmitz T. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Dec 14;377(24):2399-400. doi: 10.1056/NEJMc1713798. No abstract available. PMID 29239588
- [Background] FIGO Working Group on Good Clinical Practice in Maternal-Fetal Medicine. Good clinical practice advice: First trimester screening and prevention of pre-eclampsia in singleton pregnancy. Int J Gynaecol Obstet. 2019 Mar;144(3):325-329. doi: 10.1002/ijgo.12741. No abstract available. PMID 30710362
- [Background] Wright D, Nicolaides KH. Aspirin delays the development of preeclampsia. Am J Obstet Gynecol. 2019 Jun;220(6):580.e1-580.e6. doi: 10.1016/j.ajog.2019.02.034. Epub 2019 Feb 21. PMID 30797761